CLINICAL TRIAL: NCT01521793
Title: An Open-Label Study to Evaluate the Effects of Repeated Treatments of Oral QLT091001 on Safety and Vision Outcome in Subjects With Leber Congenital Amaurosis (LCA) or Retinitis Pigmentosa (RP) Due to Inherited Deficiencies of Retinal Pigment Epithelial 65 Protein (RPE65) or Lecithin: Retinol Acyltransferase (LRAT) (Extension of Study RET IRD 01)
Brief Title: Repeated Treatments of QLT091001 in Subjects With Leber Congenital Amaurosis or Retinitis Pigmentosa (Extension of Study RET IRD 01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RET IRD 02
Record Dates: First submitted 2012-01-06; First posted 2012-01-31 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: LCA (Leber Congenital Amaurosis); RP (Retinitis Pigmentosa)
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa | interventions — retinol acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: QLT091001 — oral QLT091001 administered once daily for 7 days

SUMMARY:
The purpose of this study is:

* To evaluate the safety of up to 3 additional courses of oral QLT091001 administered once daily for 7 days in subjects treated previously with a single 7-day course of QLT091001 in Study RET IRD 01
* To evaluate whether up to 3 additional courses of oral QLT091001 administered once daily for 7 days can maintain or improve visual function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with LCA or RP due to RPE65 or LRAT deficiency who received a 7-day treatment course of QLT091001 and completed the Day 30 visit in Study RET IRD 01
* Subjects who meet any one of the following criteria at least 1 month after start of the 7-day treatment course in Study RET IRD 01:

  * no increase in GVF (in at least 1 eye): Follow-up GVF increased ≤20% from baseline or
  * decrease in GVF (in at least 1 eye): Follow-up GVF decreased below the highest previous response by ˃20% or
  * Considered a reasonable candidate for retreatment, based on the Investigator's discretion, in consultation with the independent DSMB and the Sponsor, based on regression or lack of response in other parameters of visual function (e.g., subjective reports of changes in color vision or adaptation to low light) but who do not meet other (GVF) criteria for study entry

Exclusion Criteria:

* Subjects with any clinically important abnormal physical finding at Screening.
* Subjects who have taken any prescription or investigational oral retinoid medication (e.g., Accutane,® Soriatane®) within 6 months of Day 0 and subjects who did not tolerate their previous oral retinoid medication will be excluded regardless of the time of last exposure.
* Subjects with liver failure, uncontrolled thyroid disease, hypersensitivity to retinoids, or hypervitaminosis A
* Subjects who have taken any supplements containing ≥10,000 IU vitamin A within 60 days of screening

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Visual field | 12 months

SECONDARY OUTCOMES:
Safety will be assessed by evaluating the following: adverse events, clinical laboratory tests, ECG's and vital signs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sushanta Mallick, Study Director — QLT Inc.
Locations (6):
- United States (2):
  - The Chicago Lighthouse (University of Illinois at Chicago, Pangere Center for Inherited Retinal Disease), Chicago, Illinois
  - Wilmer Eye Institute (Johns Hopkins University), Baltimore, Maryland
- Montreal Children's Hospital, McGill University Health Centre, Montreal, Quebec, Canada
- Institute for Ophthalmic Research, University of Tubingen, Tübingen, Germany
- The Rotterdam Eye Hospital, Rotterdam, Netherlands
- Moorefield Eye Hospital, London, United Kingdom